CLINICAL TRIAL: NCT06986317
Title: Effectiveness of Positional Release Techniques and Graston Technique In Trapezius Trigger Point
Brief Title: Effectiveness of Positional Release Techniques and Graston Technique In Trigger Point
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-GCUF-079318
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Trigger point; Trapezius; Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain

STUDY DESIGN:
Intervention Model Description: This is interventional study.There are 2 groups in this study . One group will be treated with positional release techniques and second group will be treated with graston technique
Masking Description: Randomized clinical trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- positional release technique (Experimental): Positional release techniques along with therapeutic exercises
  Interventions: Other: Positional release techniques
- graston technique (Active Comparator): Graston technique along with therapeutic exercises
  Interventions: Other: Graston technique

INTERVENTIONS:
Other: Positional release techniques — Positional release techniques apply for 90 second with the frequency of 3. This protocol will given 2 times in a week.
  Arms: positional release technique
Other: Graston technique — Graston technique will apply at 45 degree to muscle fiber for 60 sec with the frequency of three. 2 session will be given per week
  Arms: graston technique

SUMMARY:
The purpose of the study is to evaluate comparative effectiveness of positional release techniques and graston technique In trapezius trigger point

ELIGIBILITY:
Inclusion Criteria:

Male and Female

Age group 18-55 years

At least one trigger point

Exclusion Criteria:

* Radiculopathy
* History of head and upper back trauma or surgery
* Tendency to hemorrhage
* Systemic disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-07-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 0 week, 1st week, 3rd week
  Used to measure neck pain, 10 is the worst possible pain and 0 means no pain.
Neck Disability Index | 0 week, 1st week, 3rd week
  Used to assess trigger point related neck related disability

SECONDARY OUTCOMES:
Goniometer | 0 week, 1st week, 3rd week
  Used to assess Cervical Range of Motion at baseline, 1st week and 3rd week

CONTACTS AND LOCATIONS:
Overall Officials: Rukhma Mauzzam, Principal Investigator — Elite College of Management Science
Locations (1):
- • Al- Raee Hospital Gujranwala • Civil Hospital Gujranwala • Elite college of Management Sciences Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalid, M., et al. (2023).
- [Background] Haq, K. and H. Riaz (2022).
- [Background] Cheatham SW, Lee M, Cain M, Baker R. The efficacy of instrument assisted soft tissue mobilization: a systematic review. J Can Chiropr Assoc. 2016 Sep;60(3):200-211. PMID 27713575
- [Background] Bethers AH, Swanson DC, Sponbeck JK, Mitchell UH, Draper DO, Feland JB, Johnson AW. Positional release therapy and therapeutic massage reduce muscle trigger and tender points. J Bodyw Mov Ther. 2021 Oct;28:264-270. doi: 10.1016/j.jbmt.2021.07.005. Epub 2021 Jul 14. PMID 34776151
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Anesthesiol Clin. 2007 Dec;25(4):841-51, vii-iii. doi: 10.1016/j.anclin.2007.07.003. PMID 18054148
- [Background] Bron C, Dommerholt JD. Etiology of myofascial trigger points. Curr Pain Headache Rep. 2012 Oct;16(5):439-44. doi: 10.1007/s11916-012-0289-4. PMID 22836591